CLINICAL TRIAL: NCT03950583
Title: The Clinical Course of Interstitial Pneumonia With Autoimmune Features: an Observational, Prospective Cohort Study
Brief Title: The Clinical Course of Interstitial Pneumonia With Autoimmune Features
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Western University, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 6476
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Interstitial Pneumonia
Keywords: interstitial lung disease; interstitial pneumonia; connective tissue disease; clinical course
MeSH Terms: conditions — Lung Diseases, Interstitial; Connective Tissue Diseases; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Interstitial pneumonia with autoimmune features (IPAF) is a chronic interstitial lung disease (ILD) with some laboratoristic and/or clinical features of autoimmune disease, but without meeting criteria of connective tissue disease (CTD), and with no other causes of ILD. Despite recent efforts to standardize the diagnosis of IPAF, subjects with IPAF represent a very heterogenous group of patients, whose prognosis and clinical course are far from being clear. It also remains to be clarified what proportion of IPAF patients develop clear features of CTD over time.

The aim of this observational trial is to define the clinical course of patients newly diagnosed with IPAF by prospectively following them for a period of 3 years, at 6-month intervals. The primary outcome will be 3-year lung transplant-free survival. The secondary outcome will be the proportion of patients who develop clinical and laboratoristic features clearly meeting criteria for a diagnosis of CTD at 3 years from the time of diagnosis of IPAF. Predictors of survival will also be studied.

DETAILED DESCRIPTION:
Objective of the study The objective of this study is to investigate the clinical course of IPAF to clarify the prognosis of this condition and to clarify the proportion of patients who develop clear clinical features of CTD over time. Patients will be followed prospectively for a period of 3 years, or until death or lung transplant (LTx). Predictors of LTx-free survival will be studied as well.

Rationale Interstitial pneumonia with autoimmune features (IPAF) is a chronic interstitial lung disease (ILD) with some laboratoristic and/or clinical features of autoimmune disease, but without meeting criteria of connective tissue disease (CTD), and with no other causes of ILD.

It is not uncommon for the interstitial pneumonia to be the first, and possibly the sole, manifestation of an otherwise occult CTD. The current international guidelines for the diagnosis of IIP recommend excluding CTD. For this reason, many cases of ILD with autoimmune features, but not fully meeting criteria for CTD, have been identified. Patients with IPAF, with the current diagnostic criteria, actually represent a sizable proportion of patients with ILD. However, the clinical course, prognosis and treatment approach to these patients remain unclear.

Despite recent efforts to standardize the diagnosis of IPAF, subjects with IPAF represent a very heterogenous group of patients, whose prognosis and clinical course are far from being clear. While the average age of diagnosis is higher than in CTD, there is still a female predominance. An autoimmune "flavor" may not necessarily mean a real autoimmune etiology, but currently the distinction is challenging. From this perspective, a multi-disciplinary approach together with Rheumatologist is particularly important. It also remains to be clarified what proportion of IPAF patients develop clear features of CTD over time. One issue for example is represented by the fact patient with IPAF may be treated with immunosuppressive agents, which may permanently mask the development of systemic features of CTD.

A clear distinction between IPAF and idiopathic pulmonary fibrosis (IPF), one of the most common types of ILD, is at the same time challenging and essential, as treatment is radically different in the two conditions. CTD and IPAF patients can definitely present with the same morphologic (radiographic or pathologic) pattern of usual interstitial pneumonia. However, patients with IPF respond to anti-fibrotic treatment, which is expensive, while patients with ILD secondary to CTD respond to immunosuppressive treatment. From a prognostic point of view, the survival of IPF is considered one of the worst among all types of ILD.

There is tendency to treat patients with IPAF with immunosuppressive therapy, but the rational for this remains unclear, given that the natural history of IPAF is not well known. One retrospective study suggested that the short-term prognosis of IPAF is better than that of IPF. Another retrospective study however showed that survival is worse than in CTD-ILD. At the same time, the latter study showed that patients with IPAF and UIP morphologic pattern had the same, poor prognosis of IPF patients, raising concern that they were actually IPF patients to start with and that they were mislabelled as IPAF. Again, the retrospective nature of these studies makes the results more difficult to interpret.

In 2015, in an effort to standardize the diagnosis of IPAF, the European Respiratory Society (ERS) and the American thoracic Society (ATS) published a research statement that outlined the proposed diagnostic criteria for IPAF. These include:

1. Presence of an interstitial pneumonia (HRCT or SLB) and,
2. Exclusion of alternative etiologies and,
3. Does not meet criteria of defined CTD and,
4. At least one feature from at least two of these domains A. Clinical Domain B. Serologic Domain C. Morphologic Domain

A. Clinical domain:

* Distal digital fissuring (i.e. "mechanic hands")
* Distal digital tip ulceration
* Inflammatory arthritis or polyarticular morning joint stiffness ≥60 min
* Palmar telangiectasia
* Raynaud's phenomenon
* Unexplained digital edema
* Unexplained fixed rash on the digital extensor surfaces (Gottron's sign)

Symptoms or signs of peripheral joint synovitis considered as evidence for inflammatory arthritis, but joint pain alone is not included due to its lack of specificity.

Other non-specific features, such as alopecia, photosensitivity, oral ulcers, weight loss, sicca symptoms, myalgia or arthralgia, are not included.

Demographic profiles that may be more frequently encountered in CTD (such as younger age and female, sex) are not included given their lack of specificity for CTD-ILD.

Digital fissuring ("mechanic hands"), Gottron's sign usually suggestive of anti-synthetase syndrome or systemic sclerosis-myositis overlap Raynaud's phenomenon, palmar telangiectasia, distal digital tip ulceration and digital edema are usually suggestive of scleroderma.

B. Serologic domain:

* ANA ≥1:320 titre, diffuse, speckled, homogeneous patterns or
* ANA nucleolar pattern (any titre) or
* ANA centromere pattern (any titre)
* Rheumatoid factor ≥2× upper limit of normal
* Anti-CCP
* Anti-dsDNA
* Anti-Ro (SS-A)
* Anti-La (SS-B)
* Anti-ribonucleoprotein
* Anti-Smith
* Anti-topoisomerase (Scl-70)
* Anti-tRNA synthetase
* Anti-PM-Scl
* Anti-MDA-5

C. Morphologic domain

* Suggestive radiology patterns by HRCT :

  1. NSIP
  2. OP
  3. NSIP with OP overlap
  4. LIP
* Histopathology patterns or features by surgical lung biopsy:

  1. NSIP
  2. OP
  3. NSIP with OP overlap
  4. LIP
  5. Interstitial lymphoid aggregates with germinal centres
* Diffuse lymphoplasmacytic infiltration (with or without lymphoid follicles)
* Multi-compartment involvement (in addition to interstitial pneumonia):

  1. Unexplained pleural effusion or thickening, pericardial effusion /thickening, intrinsic airways disease (by PFT, imaging or pathology) or pulmonary vasculopathy.

The conclusion of the research statement from ERS/ATS was that "prospective studies are urgently needed to validate the proposed classification criteria and to determine the natural history and clinical implications of a classification of IPAF", which is the purpose of this study.

Hypothesis We hypothesize that LTx-free survival in IPAF is better than in IPF, and similar to that of ILD secondary to CTD. It is also possible that different phenotypes of IPAF exist, and it may be prognostically relevant to distinguish them at the time of diagnosis.

We also hypothesize that a sizable proportion of IPAF patients may develop clear clinical or serologic features of CTD during the observation period.

ELIGIBILITY:
Inclusion Criteria:

* new diagnosis of IPAF based on the A,B,C) ERS/ATS criteria (Eur Respir J 2015;46:976-87)

Exclusion Criteria:

* Interstitial lung disease other than IPAF
* Not a new diagnosis of IPAF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a new diagnosis of interstitial pneumonia with autoimmune features, according to ERS/ATS A,B,C criteria
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Survival | 3 years
  Survival rate since the time of diagnosis

SECONDARY OUTCOMES:
Rate of development of autoimmune disease | 3 years
  Incidence of a new diagnosis of autoimmune disease during the 3-year clinical course
Clinical progression | 3 years
  Time to either: decline of FVC >10% pred; decline of 6-min walk distance >50 m; hospitalization for respiratory causes; lung transplant assessment; or death.
Acute exacerbation | 3 years
  Incidence of acute exacerbations since the time of diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Marco Mura, MD, PhD, Principal Investigator — Lawson Research Institute; Pari Basharat, MD, Principal Investigator — Lawson Research Institute
Locations (1):
- London Health Science Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fischer A, Antoniou KM, Brown KK, Cadranel J, Corte TJ, du Bois RM, Lee JS, Leslie KO, Lynch DA, Matteson EL, Mosca M, Noth I, Richeldi L, Strek ME, Swigris JJ, Wells AU, West SG, Collard HR, Cottin V; "ERS/ATS Task Force on Undifferentiated Forms of CTD-ILD". An official European Respiratory Society/American Thoracic Society research statement: interstitial pneumonia with autoimmune features. Eur Respir J. 2015 Oct;46(4):976-87. doi: 10.1183/13993003.00150-2015. Epub 2015 Jul 9. PMID 26160873
- [Result] Oldham JM, Adegunsoye A, Valenzi E, Lee C, Witt L, Chen L, Husain AN, Montner S, Chung JH, Cottin V, Fischer A, Noth I, Vij R, Strek ME. Characterisation of patients with interstitial pneumonia with autoimmune features. Eur Respir J. 2016 Jun;47(6):1767-75. doi: 10.1183/13993003.01565-2015. Epub 2016 Apr 21. PMID 27103387
- [Result] Ahmad K, Barba T, Gamondes D, Ginoux M, Khouatra C, Spagnolo P, Strek M, Thivolet-Bejui F, Traclet J, Cottin V. Interstitial pneumonia with autoimmune features: Clinical, radiologic, and histological characteristics and outcome in a series of 57 patients. Respir Med. 2017 Feb;123:56-62. doi: 10.1016/j.rmed.2016.10.017. Epub 2016 Oct 31. PMID 28137497
- [Result] Kelly BT, Moua T. Overlap of interstitial pneumonia with autoimmune features with undifferentiated connective tissue disease and contribution of UIP to mortality. Respirology. 2018 Jun;23(6):600-605. doi: 10.1111/resp.13254. Epub 2018 Jan 10. PMID 29320807
- [Result] Collins BF, Spiekerman CF, Shaw MA, Ho LA, Hayes J, Spada CA, Stamato CM, Raghu G. Idiopathic Interstitial Pneumonia Associated With Autoantibodies: A Large Case Series Followed Over 1 Year. Chest. 2017 Jul;152(1):103-112. doi: 10.1016/j.chest.2017.03.004. Epub 2017 Mar 12. PMID 28300570
- [Result] Ferri C, Manfredi A, Sebastiani M, Colaci M, Giuggioli D, Vacchi C, Della Casa G, Cerri S, Torricelli P, Luppi F. Interstitial pneumonia with autoimmune features and undifferentiated connective tissue disease: Our interdisciplinary rheumatology-pneumology experience, and review of the literature. Autoimmun Rev. 2016 Jan;15(1):61-70. doi: 10.1016/j.autrev.2015.09.003. Epub 2015 Sep 16. PMID 26384526